CLINICAL TRIAL: NCT04051684
Title: Transverse Abdominal Plane Blocks for Bariatric Surgery Patients: A Single Blinded Randomized Controlled Study
Brief Title: Regional TAP Block for Bariatric Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Karina Gritsenko, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-01-013
Record Dates: First submitted 2018-11-19; First posted 2019-08-09 (Actual); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Bariatric Surgery; Transverse Abdominal Plane Regional Blocks
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- TAP, Bupivacaine (Experimental): This group will receive general anesthesia and at the end of the operation, but still in the operating room, a single shot TAP block with 0.5% ropivacaine 15-20 ml / side under ultrasound guided technique with blunt tipped, 21 gauge needle.
  Interventions: Procedure: Transverse abdominal plane block; Drug: Ropivacaine
- No intervention (No Intervention): General anesthesia

INTERVENTIONS:
Procedure: Transverse abdominal plane block — Regional anesthesia team will perform a single shot TAP block with 0.5% ropivacaine 15-20 ml / side under ultrasound guided technique with blunt tipped, 21 gauge needle.
  Other Names: TAP
  Arms: TAP, Bupivacaine
Drug: Ropivacaine — Regional anesthesia team will perform a single shot TAP block with 0.5% ropivacaine 15-20 ml / side under ultrasound guided technique with blunt tipped, 21 gauge needle.
  Arms: TAP, Bupivacaine

SUMMARY:
Addition of transverse abdominis plane (TAP) block to general anesthesia for morbidly obese patients (BMI >35) undergoing laparoscopic bariatric surgery for weight loss will significantly reduce opioid use in the recovery room

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be 18 years of age or older and able to provide his or her own consent.
2. The patient is scheduled for bariatric surgery including laparoscopic gastric banding, sleeve gastrectomy, and gastric bypass.
3. The patient must be surgically and medically accepted for the procedure
4. Good functional status, ability to perform activities of daily living
5. The patients BMI > 35, no upper limit
6. Signed study specific informed consent prior to enrollment

Exclusion Criteria:

1. Patients with an allergy to local anesthetics
2. Patients diagnosed with peripheral neuropathies including diabetes mellitus.
3. Patients with BMI <35
4. Patients with significant coronary artery disease
5. Patient refusal of block procedure.
6. Patients with chronic pain
7. Patients on pre-operative maintenance narcotics
8. American Society of Anesthesiologist classification system 4 (ASA 4) patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Gritsenko, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP, Bupivacaine | No Intervention
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP, Bupivacaine | No Intervention | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43.5 [32.5 to 51.2] | 43 [36 to 53] | 43.5 [35 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Opioid Usage
Description: The amounts of opioids used by the patient will be collected by a person blinded to the allocation group
Time Frame: 24 hour after surgery
Measure: Median (Inter-Quartile Range); unit: morphine equivalent
Arm/Group | TAP, Bupivacaine | No Intervention
Number analyzed (Participants) | 12 | 11
morphine equivalent | 2.25 [2.25 to 4] | 4 [2 to 4]

2. Secondary Outcome: Pain Score Assessed With Visual Analog Score (VAS)
Description: Visual Analog Score (VAS) scores correlate to Pain scores (0-10, 0 being no pain and 10 being the worst pain). VAS will be taken within 30 minutes of arrival to post anesthesia care unit (PACU)
Time Frame: 30 minutes within arrival to PACU
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAP, Bupivacaine | No Intervention
Number analyzed (Participants) | 12 | 11
units on a scale | 5.5 [4.25 to 8.25] | 2 [1 to 3]

3. Secondary Outcome: Nausea: The Number of Participants Experiencing Nausea Will be Assessed by Chart Review
Description: The number of participants experiencing nausea will be assessed by chart review
Time Frame: Up to 5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | TAP, Bupivacaine | No Intervention
Number analyzed (Participants) | 12 | 11
Participants | 5 | 3

4. Secondary Outcome: Vomiting: The Number of Participants Experiencing Vomiting Will be Assessed by Chart Review
Description: The number of participants experiencing vomiting will be assessed by chart review
Time Frame: Up to 5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | TAP, Bupivacaine | No Intervention
Number analyzed (Participants) | 12 | 11
Participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | TAP, Bupivacaine | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes